CLINICAL TRIAL: NCT04367129
Title: Electrocardiogram Analysis in COVID-19 Patients
Acronym: ELCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Other Study IDs: 385/2020/Oss/AOUFe
Record Dates: First submitted 2020-04-16; First posted 2020-04-29 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-04

CONDITIONS: SARS-CoV Infection
Keywords: ECG; SARS-CoV-2 Infection; Mortality; Invasive mechanical ventilation
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ECG — 12 lead electrocardiogram

SUMMARY:
Electrocardiographic (ECG) evaluation of patients with severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2) infection.

The present study involves three different phases of evaluation of the ECG traces of hospitalized patients with SARS-CoV-2 infection.

* Phase 1: it is proposed to collect and retrospectively analyze the ECGs of hospitalized patients with severe SARS-CoV-2 infection which led to invasive ventilation or patient death as a consequence and, if available, also possible troponin dosage;
* Phase 2: aims to collect and analyze the ECGs of consecutive hospitalized patients with SARS-CoV-2 infection and evaluate their relationship with the course of the disease, cardiac involvement and prognosis;
* Phase 3: it is proposed to repeat ECG and to carry out echocardiogram to patients with SARS-CoV-2 infection after 3 months from hospital discharge by simultaneously performing, if deemed clinically indicated, also cardiac magnetic resonance. In this phase, any evolutions of ECG alterations of the acute phase will be described and the relationship with cardiac involvement will be assessed.

DETAILED DESCRIPTION:
In the early months of 2020, SARS-CoV-2 virus infection quickly spread around the world to a pandemic. On 2 April 2020, confirmed cases of coronavirus disease 2019 (COVID-19) worldwide exceeded one million and an unprecedented health crisis has occurred in recent history.

SARS-CoV-2 disease can lead to the development of even severe pneumonia with the need for ventilatory support and in some cases fatal outcome.

From the data currently present in the literature, important relationships emerge between infection and cardiovascular diseases. COVID-19 patients with underlying pre-existing heart disease or cardiovascular risk factors have a more severe course of the disease and are more at risk of adverse outcomes and death than individuals with no history of heart disease or risk factors.

During the course of the infection, some patients even without previous heart disease may experience myocardial injury and this leads to a significant increase in in-hospital mortality. Myocardial pain during SARS-CoV-2 infection is associated with cardiac dysfunction and arrhythmias.

To date, there are no data on the role of the electrocardiogram neither in the diagnosis of cardiac involvement nor in predicting the prognosis of patients with SARS-CoV-2 infection.

Whether there are basal electrocardiographic features capable of correlating with the course of the disease and the prognosis is currently unknown. The development of electrocardiographic changes during the course of the disease and their possible prognostic significance has not currently been described.

The present study involves three different phases of evaluation of the electrocardiographic (ECG) traces of hospitalized patients with SARS-CoV-2 infection.

* Phase 1: it is proposed to collect and retrospectively analyze the ECGs of hospitalized patients with severe SARS-CoV-2 infection which led to invasive ventilation or patient death as a consequence and, if available, also possible troponin dosage;
* Phase 2: aims to collect and analyze the ECGs of consecutive hospitalized patients with SARS-CoV-2 infection and evaluate their relationship with the course of the disease, cardiac involvement and prognosis;
* Phase 3: it is proposed to repeat ECG and to carry out echocardiogram to patients with SARS-CoV-2 infection after 3 months from hospital discharge by simultaneously performing, if deemed clinically indicated, also cardiac magnetic resonance. In this phase, any evolutions of ECG alterations of the acute phase will be described and the relationship with cardiac involvement will be assessed.

Phase 1 Retrospective, multicentric, cohort study Phase 2 and 3 prospective, multicentric, cohort study

Phase 1:

• Describe the ECG characteristics in patients presenting with severe form of SARS-CoV-2 infection

Phase 2:

* To evaluate the correlation between ECG signs and cardiac involvement in the acute phase
* Assess the correlation between ECG signs and mortality/invasive mechanical ventilation in the acute phase secondary:
* To evaluate the prevalence of ECG changes in the enrolled population
* Analyze the prevalence of various cardiovascular risk factors in the enrolled population
* Examine the impact of ECG changes on the short-term prognosis
* Explore new possible prognostic risk factors

Phase 3:

* To evaluate the correlation between acute phase ECG signs and chronic phase cardiac involvement
* To evaluate the appearance, in the short-term follow-up, of signs of cardiac involvement (cardiomyopathies and conduction disorders in particular)

Data collected:

* demographic characteristics
* cardiovascular risk factors
* comorbidities
* blood tests including cardiac markers (troponin, BNP) collected in multiple points if available
* radiographic examinations and echocardiogram (if performed)
* ECG traces performed at onset, worsening and / or troponin peak
* length of hospital stay
* treatments administered
* complications
* clinical outcome

Enrolled patients will be followed clinically until the day of discharge as per care practice. A 3-month follow-up is foreseen to evaluate the outcome and repeat the ECG. At the discretion of the clinician who manages the patient, transthoracic echocardiogram and / or cardiac magnetic resonance imaging will also be performed.

A formal calculation of the sample size is not possible due to the total lack of data. Furthermore, since it is an observational project, the calculation of the sample size is not mandatory. However, based on similar studies, it is believed that the minimum samples for the various phases are:

80 patients for Phase 1 study objectives, 800 patients for Phase 2 study objectives and 300 patients for Phase 3 study objectives

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old
* confirmed SARS-CoV-2 infection (pharyngeal swab positive for viral RNA or clinical diagnosis of COVID-19 based on chest x-ray or high resolution CT)
* hospitalization in a hospital setting

Exclusion Criteria:

* SARS-CoV-2 infection not confirmed by pharyngeal swab or clinical-radiographic criteria
* absence of ECG tracing performed at the time of hospitalization

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 1014 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: ECG characteristics in patients presenting with severe form of SARS-CoV-2 infection | 1 month
  Describe the ECG characteristics in patients presenting with severe form of SARS-CoV-2 infection
Phase 2: Correlation between ECG signs and needs for invasive mechanical ventilation and/or mortality in the acute phase | 6 months
  To evaluate the correlation between ECG signs and cardiac involvement in the acute phase
  • Assess the correlation between ECG signs and mortality in the acute phase
Phase 3: Correlation between ECG signs and cardiac involvement and mortality in the chronic phase | 12 months
  To evaluate the correlation between acute phase ECG signs and chronic phase cardiac involvement
  • evaluate the appearance, in the short-term follow-up, of signs of cardiac involvement (cardiomyopathies and conduction disorders in particular)

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Bertini, MD, PhD, Principal Investigator — s.anna university hospital
Locations (1):
- Arcispedale S. Anna, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided a plan to share individual participant data (IPD)

REFERENCES:
- [Background] Bonow RO, Fonarow GC, O'Gara PT, Yancy CW. Association of Coronavirus Disease 2019 (COVID-19) With Myocardial Injury and Mortality. JAMA Cardiol. 2020 Jul 1;5(7):751-753. doi: 10.1001/jamacardio.2020.1105. No abstract available. PMID 32219362
- [Background] Guo T, Fan Y, Chen M, Wu X, Zhang L, He T, Wang H, Wan J, Wang X, Lu Z. Cardiovascular Implications of Fatal Outcomes of Patients With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):811-818. doi: 10.1001/jamacardio.2020.1017. PMID 32219356
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Derived] Zuin M, Ferrari R, Guardigli G, Malagu M, Vitali F, Zucchetti O, D'Aniello E, Di Ienno L, Gibiino F, Cimaglia P, Grosseto D, Corzani A, Galvani M, Ortolani P, Rubboli A, Tortorici G, Casella G, Sassone B, Navazio A, Rossi L, Aschieri D, Mezzanotte R, Manfrini M, Bertini M. A COVID-19 specific multiparametric and ECG-based score for the prediction of in-hospital mortality: ELCOVID score. Intern Emerg Med. 2024 Aug;19(5):1279-1290. doi: 10.1007/s11739-024-03599-3. Epub 2024 Apr 23. PMID 38652232
- [Derived] Bertini M, Ferrari R, Guardigli G, Malagu M, Vitali F, Zucchetti O, D'Aniello E, Volta CA, Cimaglia P, Piovaccari G, Corzani A, Galvani M, Ortolani P, Rubboli A, Tortorici G, Casella G, Sassone B, Navazio A, Rossi L, Aschieri D, Rapezzi C. Electrocardiographic features of 431 consecutive, critically ill COVID-19 patients: an insight into the mechanisms of cardiac involvement. Europace. 2020 Dec 23;22(12):1848-1854. doi: 10.1093/europace/euaa258. PMID 32944767